CLINICAL TRIAL: NCT03517319
Title: Dose-response Relationship of Botullinum Toxin (DWP 450) for Finger Flexor Spasticity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Shi-Uk Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 26-2016-103
Record Dates: First submitted 2018-04-17; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Spasticity as Sequela of Stroke
MeSH Terms: interventions — Saline Solution; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Normal Saline 0.9% 1.2 ml will be injected to finger flexor muscles
  Interventions: Drug: Normal Saline 0.9% 1.2 ml
- Treatment dose 15 (Experimental): Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 15 U will be injected to finger flexor muscles
  Interventions: Drug: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 15 U
- Treatment dose 30 (Experimental): Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 30 U will be injected to finger flexor muscles
  Interventions: Drug: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 30 U
- Treatment dose 50 (Experimental): Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 50 U will be injected to finger flexor muscles
  Interventions: Drug: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 50 U
- Treatment dose 70 (Experimental): Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 70 U will be injected to finger flexor muscles
  Interventions: Drug: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 70 U

INTERVENTIONS:
Drug: Normal Saline 0.9% 1.2 ml
  Arms: Placebo
Drug: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 15 U
  Other Names: Nabota (DWP 450)
  Arms: Treatment dose 15
Drug: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 30 U
  Other Names: Nabota (DWP 450)
  Arms: Treatment dose 30
Drug: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 50 U
  Other Names: Nabota (DWP 450)
  Arms: Treatment dose 50
Drug: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 70 U
  Other Names: Nabota (DWP 450)
  Arms: Treatment dose 70

SUMMARY:
Study Design: Randomized Single Blind Study Objective: To determine the dose relationship of DWP 450 for finger flexor spasticity Subjects: 78 patients with upper extremity spasticity after CVA Inclusion criteria: Patient who have spasticity (MAS greater than 2 in finger flexors) Methods: Patients will be randomly assigned to one of 5 groups. Gp 1: placebo, Gp 2: 15U, Gp 3: 30 U, Gp 4: 50 U, Gp 5: 75 U

DETAILED DESCRIPTION:
Seventy-eight patients with upper extremity spasticity after cerebrovascular accident will be recruited and randomly assigned to one of 5 groups. The groups are as followings.

Gp 1: placebo group (Normal saline 1.2 ml) Gp 2: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 15 U Gp 3: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 30 U Gp 4: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 50 U Gp 5: Clostridium Botulinum Toxin Type A (Nabota, DWP 450) 70 U

According to the group, the injection will be performed to the finger flexor musles (flexor digitorum superficialis and profundus). Outcome measurement will be MAS (Modified ashworth scale), FMA, Wolf Motor Assessment, Cross sectional area measured by Ultrasonography.

Patient evaluation will be conducted 2 weeks, 1 months, 2 months, and 3 months after the injection.

ELIGIBILITY:
Inclusion Criteria:

* over 6 weeks after stroke onset
* MAS (modified Ashworth scale) greater than 2 in finger flexor

Exclusion Criteria:

* neuromuscular junction disease or motor neuron disease
* phenol or alcohol block for the target limbs within 6 months before screening
* botulinum toxin injection within 3 months before screening
* history or plan for tendon lengthening surgery
* significant contracture ormuscle atrophy at the target joint or muscle
* concurrent treatment with intrathecal baclofen
* hypersensitivity or allergy to study drug or its components
* pregnancy or planned pregnancy, breastfeeding
* abnormal lab findings for alanine aminotransferase, aspartate aminotransferase, blood urea nitrogen, and serum creatinine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
MAS (Modified Ashworth Scale) | baseline
  Spasticity measurement measures resistance during passive soft-tissue stretching(taken from Bohannon and Smith, 1987):
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
MAS (Modified Ashworth Scale) | 2wks after injection
  Spasticity measurement measures resistance during passive soft-tissue stretching(taken from Bohannon and Smith, 1987):
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
MAS (Modified Ashworth Scale) | 4wks after injection
  Spasticity measurement measures resistance during passive soft-tissue stretching(taken from Bohannon and Smith, 1987):
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
MAS (Modified Ashworth Scale) | 8wks after injection
  Spasticity measurement measures resistance during passive soft-tissue stretching(taken from Bohannon and Smith, 1987):
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
MAS (Modified Ashworth Scale) | 12wks after injection
  Spasticity measurement measures resistance during passive soft-tissue stretching(taken from Bohannon and Smith, 1987):
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension

SECONDARY OUTCOMES:
Ultrasonography | baseline
  measurement of changes of cross sectional area
Ultrasonography | 2wks after injection
  measurement of changes of cross sectional area
Ultrasonography | 4wks after injection
  measurement of changes of cross sectional area
Ultrasonography | 8wks after injection
  measurement of changes of cross sectional area
Ultrasonography | 12wks after injection
  measurement of changes of cross sectional area
Fugl Myer Upper Extremity Assessment | baseline
  measurement of upper extremity function
Fugl Myer Upper Extremity Assessment | 2 wks after injection
  measurement of upper extremity function
Fugl Myer Upper Extremity Assessment | 4 wks after injection
  measurement of upper extremity function
Fugl Myer Upper Extremity Assessment | 8 wks after injection
  measurement of upper extremity function
Fugl Myer Upper Extremity Assessment | 12 wks after injection
  measurement of upper extremity function
Wolf Motor Assessment | baseline
  measurement of upper extremity function
Wolf Motor Assessment | 2 wks after injection
  measurement of upper extremity function
Wolf Motor Assessment | 4 wks after injection
  measurement of upper extremity function
Wolf Motor Assessment | 8 wks after injection
  measurement of upper extremity function
Wolf Motor Assessment | 12 wks after injection
  measurement of upper extremity function

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Uk Lee, Study Chair — Seoul National University
Locations (1):
- Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Seoul, Dong Jak Ku, South Korea

IPD SHARING:
Plan to Share IPD: No